CLINICAL TRIAL: NCT02722109
Title: Dual Energy CT: A New Method for Better Dose Calculation in Proton Beam Therapy
Acronym: (DUAL)
Status: Terminated | Type: Observational
Why Stopped: Not enough patients signed up
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Vicki Trier Taasti, M.Sc., PhD student, Aarhus University Hospital
Other Study IDs: VEK52217
Record Dates: First submitted 2016-03-15; First posted 2016-03-29 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention will be done

SUMMARY:
Researchers want to compare proton stopping ratios, used for proton beam therapy planning, calculated based on single energy CT and dual energy CT images; with the intension of improve upon the proton range determination.

DETAILED DESCRIPTION:
The main goal of this study is to compare proton stopping ratios, used for proton beam therapy planning, calculated based on single energy CT and dual energy CT images.

The calculation methods for proton stopping power ratios differs for the two types of CT images, and researchers want to investigate if the proton stopping power ratio can be estimated more accurately by using dual energy CT. A more accurate stopping power ratio calculation gives a more accurate proton range determination in the patient tissue, which again will lead to a better knowledge of the dose distribution in the patient undergoing cancer treatment with proton beam irradiation.

Knowing the accurate dose distribution allows for an uncertainty margin reduction around the tumor, which will result in less normal tissue being irradiated and thereby the risk of side effects is reduced without risking an under-dosage of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who are scheduled for a control CT scan

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with a identified tumor referred to curativ intended external beam radiotherapy
  * Patients, for who are scheduled for a control CT scan during their treatment course
  * Patients above 18 years of age
  * Participation will take place on a voluntary basis It is estimated that annually around 1,000 patients will meet the above inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Stopping power ratio differences | 2 months
  For each patient the stopping power will be calculated based on both single and dual energy CT. The treatment of the patient will not be affected in any way of this study, the patient will receive the same treatment whether or not the patient volunteers to participate in this study. And the outcome of the calculations performed in this study will have no influence for the patient.
  The calculations of the stopping power differences for each patient will as far as possible be done right after acquisition of the CT images, but the exact time point is not important. We will set as a deadline that the calculation for each patient is done within 2 months of acquisition of the CT images of the patient.
  The entire study will be finished within 2 years, and the results will be tried published in a peer-reviewed journal.

CONTACTS AND LOCATIONS:
Overall Officials: Cai Grau, Professor, Study Director — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other centers

REFERENCES:
- [Background] Engelsman M, Schwarz M, Dong L. Physics controversies in proton therapy. Semin Radiat Oncol. 2013 Apr;23(2):88-96. doi: 10.1016/j.semradonc.2012.11.003. PMID 23473685
- [Background] Knopf AC, Lomax A. In vivo proton range verification: a review. Phys Med Biol. 2013 Aug 7;58(15):R131-60. doi: 10.1088/0031-9155/58/15/R131. Epub 2013 Jul 17. PMID 23863203
- [Background] Johnson TR. Dual-energy CT: general principles. AJR Am J Roentgenol. 2012 Nov;199(5 Suppl):S3-8. doi: 10.2214/AJR.12.9116. PMID 23097165
- [Background] Hunemohr N, Krauss B, Tremmel C, Ackermann B, Jakel O, Greilich S. Experimental verification of ion stopping power prediction from dual energy CT data in tissue surrogates. Phys Med Biol. 2014 Jan 6;59(1):83-96. doi: 10.1088/0031-9155/59/1/83. Epub 2013 Dec 12. PMID 24334601
- [Background] Bourque AE, Carrier JF, Bouchard H. A stoichiometric calibration method for dual energy computed tomography. Phys Med Biol. 2014 Apr 21;59(8):2059-88. doi: 10.1088/0031-9155/59/8/2059. Epub 2014 Apr 2. PMID 24694786
- [Background] Hall EJ. Henry S. Kaplan Distinguished Scientist Award 2003. The crooked shall be made straight; dose-response relationships for carcinogenesis. Int J Radiat Biol. 2004 May;80(5):327-37. doi: 10.1080/09553000410001695895. PMID 15223765
- [Result] Paganetti H. Range uncertainties in proton therapy and the role of Monte Carlo simulations. Phys Med Biol. 2012 Jun 7;57(11):R99-117. doi: 10.1088/0031-9155/57/11/R99. Epub 2012 May 9. PMID 22571913
- [Result] Hudobivnik N, Schwarz F, Johnson T, Agolli L, Dedes G, Tessonnier T, Verhaegen F, Thieke C, Belka C, Sommer WH, Parodi K, Landry G. Comparison of proton therapy treatment planning for head tumors with a pencil beam algorithm on dual and single energy CT images. Med Phys. 2016 Jan;43(1):495. doi: 10.1118/1.4939106. PMID 26745942
- [Result] Hansen DC, Seco J, Sorensen TS, Petersen JB, Wildberger JE, Verhaegen F, Landry G. A simulation study on proton computed tomography (CT) stopping power accuracy using dual energy CT scans as benchmark. Acta Oncol. 2015;54(9):1638-42. doi: 10.3109/0284186X.2015.1061212. Epub 2015 Jul 29. PMID 26219959
- [Result] Yang M, Virshup G, Clayton J, Zhu XR, Mohan R, Dong L. Theoretical variance analysis of single- and dual-energy computed tomography methods for calculating proton stopping power ratios of biological tissues. Phys Med Biol. 2010 Mar 7;55(5):1343-62. doi: 10.1088/0031-9155/55/5/006. Epub 2010 Feb 10. PMID 20145291
- [Result] Schneider U, Pedroni E, Lomax A. The calibration of CT Hounsfield units for radiotherapy treatment planning. Phys Med Biol. 1996 Jan;41(1):111-24. doi: 10.1088/0031-9155/41/1/009. PMID 8685250